CLINICAL TRIAL: NCT01998009
Title: Performance Characteristics of Immunochemical and Guaiac FOBT
Brief Title: Study of In-home Tests for Colorectal Cancer
Acronym: SIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Battelle Memorial Institute (Other); University of Minnesota (Other); Indiana University (Other); Park Nicollet Health Services (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDC-NCCDPHP-5985
Record Dates: First submitted 2013-11-06; First posted 2013-11-28 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2015-02

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; mass screening; fecal occult blood
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal occult blood tests (Other): Each patient will perform one guaiac and two immunochemical fecal occult blood tests at home.
  Interventions: Other: fecal occult blood tests

INTERVENTIONS:
Other: fecal occult blood tests

SUMMARY:
The objective of this study is to compare the performance characteristics or accuracy of different in-home screening tests for colorectal cancer (fecal occult blood tests), among patients without symptoms of colorectal cancer. Patients who meet study eligibility criteria and agree to participate in the study are asked to perform one guaiac and two immunochemical fecal occult blood tests at home prior to their colonoscopy. After the patient has completed and sent in the test kits, the patient then undergoes their previously scheduled colonoscopy. Accuracy and performance characteristics for each type of fecal occult blood test, including sensitivity, specificity, test positivity rate and positive predictive value for advanced colorectal neoplasia (advanced colorectal polyps) or colorectal cancer, will be estimated by comparing the fecal occult blood test results with the results of the colonoscopy.

DETAILED DESCRIPTION:
One of the recommended options for colorectal cancer screening in the population at average risk for colorectal cancer is annual fecal occult blood test (FOBT) starting at age 50. Randomized controlled trials have shown that annual or biennial fecal occult blood testing using a guaiac-based test reduces incidence and mortality from colorectal cancer. However, the sensitivity and specificity of the guaiac-based tests is relatively low. Guaiac-based fecal tests can produce false-positive or false-negative results with certain foods, vitamins, or medications, so dietary restrictions are generally recommended before the test. Newer, immunochemical FOBTs use antibodies to detect the globin portion of human hemoglobin and do not require dietary restrictions. These immunochemical tests may have improved performance characteristics (sensitivity and specificity) compared with the guaiac-based tests. However, there have been few studies of the performance characteristics of the immunochemical tests in the average-risk population, particularly for the iFOBTs that are currently available in the U.S. There are several iFOBT tests on the U.S. market which may have different performance characteristics.

Some of the newer immunochemical tests also have the advantage of having a simpler sampling procedure for the patient. Guaiac-based FOBTs generally use sticks or spatulas to collect specimens from three stools that have not contacted toilet bowl water; these specimens are then smeared on test cards. However, some immunochemical tests allow sample collection by brushing the surface of the stool while it is in the toilet bowl water. In addition, some immunochemical tests only require samples from one or two stools.

Colorectal cancer is a leading cause of cancer-related morbidity and mortality. Key policy groups including the ACS, the American College of Radiology, the U.S. Multi-society Task Force on Colorectal Cancer, and the U.S. Preventive Services Task Force recommend the FOBT (guaiac or immunochemical-based) as one of several appropriate screening strategies for colorectal cancer. Although colonoscopy has higher sensitivity and specificity than FOBT in detecting advanced colorectal neoplasia, colonoscopy is an invasive test that has several potential disadvantages when screening the average-risk population, including higher costs, capacity limitations, and increased risk of complications. Immunochemical FOBT may have some advantages over both guaiac-based FOBT and colonoscopy for screening the average-risk population, including better performance characteristics and better patient acceptability than gFOBT and lower costs than colonoscopy. Unfortunately, the scientific literature on the sensitivity and specificity of the respective tests is not sufficient to support more specific recommendations about which test is best for routine screening among asymptomatic adults. This study will address that crucial gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* 50 - 75 years of age
* Scheduled to have a colonoscopy for screening or as a routine exam
* Has not had more than one episode of rectal bleeding in the last 6 months
* Does not have a personal history of colorectal cancer or colorectal polyps
* Has not had a positive FOBT in the 12 months prior to study enrollment
* Has not had a colonoscopy within the past 5 years
* Has not had a prior colon resection or colon or rectal surgery
* Does not have a history of inflammatory bowel disease (e.g. ulcerative colitis or Crohn's disease)
* Does not have a personal or family history of familial adenomatous polyposis (FAP) or hereditary nonpolyposis colorectal cancer (HNPCC)
* Not currently taking anticoagulant medication such as Coumadin, Warfarin, Heparin, or Plavix
* Able to read English

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1382 (Actual)
Dates: Start 2011-05; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with a positive colonoscopy finding indicating an advanced colorectal neoplasia who also have a positive fecal occult blood test result | at time of colonoscopy
  This outcome will assess the sensitivity of the fecal occult blood test for detection of advanced colorectal neoplasia. Advanced colorectal neoplasia will be defined as an adenoma with a diameter of 10 mm or more, a villous adenoma, a tubulovillous adenoma, an adenoma with high-grade dysplasia, carcinoma in situ, or invasive cancer. For each type of fecal occult blood test, the sensitivity for advanced colorectal neoplasia will be estimated by comparing the fecal occult blood test results with the results of the colonoscopy.

SECONDARY OUTCOMES:
The proportion of participants with a negative colonoscopy finding who also have a negative fecal occult blood test result | at time of colonoscopy
  This outcome will assess the specificity of the fecal occult blood test for detection of advanced colorectal neoplasia. Advanced colorectal neoplasia will be defined as an adenoma with a diameter of 10 mm or more, a villous adenoma, a tubulovillous adenoma, an adenoma with high-grade dysplasia, carcinoma in situ, or invasive cancer. For each type of fecal occult blood test, the specificity for advanced colorectal neoplasia will be estimated by comparing the fecal occult blood test results with the results of the colonoscopy.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota